CLINICAL TRIAL: NCT05742581
Title: Evaluation of the Relationship Between Critical Shoulder Angle and Acromial Index Measurements With Rotator Cuff Rupture on 3D Models
Brief Title: Critical Shoulder Angle and Acromial Index on 3D Models
Status: Completed | Type: Observational
Sponsor: Merve Sevgi INCE (Other)
Responsible Party: Sponsor-Investigator, Merve Sevgi INCE, Teaching Assistant, Lecturer, Yuksek Ihtisas University
Organization: Yuksek Ihtisas University (Other)
Other Study IDs: 12022023
Record Dates: First submitted 2023-02-11; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Shoulder Injuries; Rotator Cuff Tears; Rotator Cuff Injuries
MeSH Terms: conditions — Shoulder Injuries; Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The rotator cuff tear group
  Interventions: Other: Computed Tomography
- Control group
  Interventions: Other: Computed Tomography

INTERVENTIONS:
Other: Computed Tomography — In our study, computerized tomography of 24 rotator cuff tears (rotator cuff tear group) and 20 Bankart lesions, and no rotator cuff tears (control group) were examined. CSA and AI were measured on three-dimensional glenohumeral joint models obtained by three-dimensional reconstructions of computed tomography examinations.

SUMMARY:
Objective: The relationship between rotator cuff tears and morphological features of the shoulder joint has not been fully explained. The earlier studies are usually done with two-dimensional radiography images, but joint positions and bone formations could not be fully evaluated in two-dimensional images. This study aims to evaluate the relationship between rotator cuff tears and critical shoulder angle (CSA) and acromial index (AI) values in three dimensions.

Methods: This study examined computerized tomography of 24 rotator cuff tears (rotator cuff tear group) and 20 Bankart lesions, and no rotator cuff tears (control group). CSA and AI were measured on three-dimensional glenohumeral joint models obtained by three-dimensional reconstructions of computed tomography examinations.

The investigators anticipate results of this study will guide clinicians in revealing the etiology of rotator cuff degeneration and determining the surgical method to be used for treatment.

ELIGIBILITY:
Inclusion Criteria:

* A total of 44 patients, including 24 patients with proven rotator cuff tear by arthroscopic surgery (rotator cuff tear group) and 20 patients with proven Bankart lesion and no rotator cuff tear by arthroscopic surgery (control group), were included in the study.

Exclusion Criteria:

* Those with an inflammatory disease and trauma history were not included in the study.

Ages: 17 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: In this study, computed tomography examinations of patients who applied to Gazi University Faculty of Medicine Department of Orthopedics and Traumatology between 2016-2019 were examined retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Critical Shoulder Angle | 2 hours
  The critical shoulder angle is defined as the angle formed between the plane of the glenoid and the line connecting the most lateral border of the acromion process, as seen on the true anteroposterior radiograph of the shoulder.
Acromial Index | 2 hours
  The acromial index is the distance between the glenoid plane and the lateral border of the acromion divided by the distance between the glenoid plane and the lateral aspect of the humeral head.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuksek Ihtisas University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watanabe A, Ono Q, Nishigami T, Hirooka T, Machida H. Association between the Critical Shoulder Angle and Rotator Cuff Tears in Japan. Acta Med Okayama. 2018 Dec;72(6):547-551. doi: 10.18926/AMO/56371. PMID 30573908